CLINICAL TRIAL: NCT01771484
Title: Clinical Efficacy of High-Sodium Diet and External Abdominal Compression in the Treatment of Orthostatic Intolerance in POTS
Brief Title: High Sodium Diet and External Abdominal Compression in POTS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not enough volunteer recruited before funding could be secured.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 121178
Record Dates: First submitted 2012-12-12; First posted 2013-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: tachycardia; pots; orthostatic intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Tachycardia; Orthostatic Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Sodium Diet (Experimental): participants will consume a diet (10 milliequivalent Na+/day)for 4-5 days prior to study day.
  Interventions: Device: External automated abdominal binder
- High sodium diet (Experimental): Participants will consume a diet high in sodium (300 milliequivalent Na+/day) for 4-5 days prior to study intervention.
  Interventions: Device: External automated abdominal binder

INTERVENTIONS:
Device: External automated abdominal binder — Participants will wear the abdominal compression binder on day 4 or 5 of the study diet. Seated and standing vitals will be collected before and during application of binder.

SUMMARY:
The investigators will test to determine if an external Automated Abdominal Binder (non-commercial product) during high sodium diet improves orthostatic tolerance, compared to wearing the binder during a low sodium diet session.

DETAILED DESCRIPTION:
The study will involve a crossover design in which each subject will be assessed (as below) while on a very low-sodium (10 milliequivalent/day) diet compared with a very high-sodium diet (300 milliequivalent/day). These acute dietary interventions will be part of the parent study ("Dietary Salt in Postural Tachycardia Syndrome" IRB#111261) for 4-5 days at the time of the study. Dietary success will be assessed using a 24h urine for sodium and creatinine as a part of the parent study.

Study Day:

* Studies will be performed at the end of the low and high-sodium diet phases.
* Blood pressure recording will not begin until at least 2 hours after the last meal (to avoid any confounding hypotension from the last meal).
* Subject will be asked to void prior to data collection.
* The subject will be seated in a chair, with their feet comfortably on the floor.
* The Dinamap electrocardiographic and blood pressure (brachial cuff) recorder will be attached to the patient and set up for measurements every 10 minutes throughout the study with digital download into the Autonomic Dysfunction Center BP database.
* After a 20-minute seated baseline, the subject will stand for up to10 minutes. Heart rate and blood pressure (HR/BP) will be measured at 1, 3, 5, and 10 minutes of standing. At the end of the baseline stand period, subjects will be asked to rate their symptoms using the provided orthostatic intolerance Symptoms questionnaire.
* The subject will then be seated and the abdominal binder will be applied without compression.
* The Dinamap electrocardiographic and blood pressure (brachial cuff) recorder will be attached to the patient and set up for measurements every 10 minutes throughout the study with digital download into the Autonomic Dysfunction Center BP database.
* At 1 and 2 hours post intervention, the subject will be asked to stand for up to 10 minutes while applying external automated abdominal binder compression (up to 40 mmHg). HR/BP will be measured at 1, 3, 5, and 10 minutes of standing.

  o If nursing staffing shortages make q1h standing difficult, then the subject should be asked to stand at least at 2 hours post intervention.
* Study termination for that day.

ELIGIBILITY:
Inclusion Criteria:

* Postural Tachycardia Syndrome: Diagnosed with POTS by the Vanderbilt Autonomic Dysfunction Center
* Increase in heart rate ≥30 beats/min with position change from supine to standing (10 minutes)
* Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence
* Participation in the parent study "Dietary Salt in Postural Tachycardia Syndrome" (IRB#111261)
* Age between 18-60 years
* Male and females
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Inability to give, or withdrawal of, informed consent
* Pregnancy
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in orthostatic tachycardia | 2 hours post baseline
  The primary end point is the change from baseline in orthostatic heart rate (change in HR on standing from a seated position) 2 hrs after baseline.

SECONDARY OUTCOMES:
Change from baseline in orthostatic symptoms | 2 hours post baseline
  The secondary endpoint is the change from baseline in orthostatic symptoms (total score) 2 hours after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States